CLINICAL TRIAL: NCT03731117
Title: FURosemide Stress Test to Predict Need of Renal Replacement THERapy in Ischemic Acute Tubular Necrosis in ICU
Acronym: FURTHER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study end date exceeded and insufficient number of subjects needed for analysis. 11 patients included / 70 theoretical patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170404J
Record Dates: First submitted 2018-10-10; First posted 2018-11-06 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury
Keywords: Ischemic Acute Kidney Injury; Intensive care units; AKI; ICU; FST; FUROSEMIDE STRESS TEST; RRT; Renal Replacement Therapy; sepsis; Cardio-pulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury; Sepsis | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative, multicenter, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FST (Experimental): FUROSEMIDE STRESS TEST
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Furosemide (FUROSEMIDE®) 20 mg / 2ml, ampoule for injection
  1 mg / kg slow intravenous injection 1.5 mg / kg if chronic exposure to diuretics in the week prior to inclusion Measurement of urine output after two and six hours. Compensation of diuresis by same volume of crystalloids over a 6-hour period
  Other Names: furosemide stress test

SUMMARY:
Ischemic acute tubular necrosis (ATN) is one of the main cause of acute kidney injury (AKI) in intensive care units (ICU). Sepsis and cardio-pulmonary bypass (CPB) are major providers. There is no validated tool to predict the evolution of AKI is ICU. Furosemide Stress Test (FST) may predict evolution of ATN-related AKI outside ICU in terms of progressive AKI, need for renal replacement therapy (RRT) or inpatient mortality with improved performance comparing to biomarkers. FST has not been validated in a prospective cohort in ICU in the settings of ischemic ATN. FURTHER aim to determine whether FST would be a useful tool to identify patients with slight to moderate AKI (KDIGO stage 1 and 2) who will evolve towards need for RRT following AKIKI (The Artificial Kidney Initiation in Kidney Injury ) delayed initiation criteria.

DETAILED DESCRIPTION:
FURTHER will enroll consecutive patients with AKI KDIGO stage 1 or 2 associated with a sepsis or following a cardiac surgery with CPB within 72h. Patients must have achieved a hemodynamic stabilization confirmed by clinical (no need for intravenous fluids, no significant variation of noradrenaline) and non-clinical (trans-thoracic echocardiography, passive leg rise or other validated tool) assessment. Included patients will receive 1 to 1.5 mg/kg of FUROSEMIDE. Urine output will be measured for 6 hours and compensated by the same volume of intravenous crystalloids. Need for RRT will be assess at 2-hour, 6-hour and daily up to day 7, following the AKIKI-study delayed initiation arm criteria. FURTHER aim to evaluate FST in a well-defined prospective cohort of ischemic ATN-related AKI as predictor of need for RRT within a week.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Hospitalized in ICU at day of inclusion
* Diagnosis of sepsis defined as proven or suspected infection and increase of the SOFA (Sequential Organ Failure Assessment) score by 2 points or more compared to basal OR Cardiothoracic surgery with CBP (Cardiopulmonary bypass) within 72 hours before inclusion
* Adequate cardiac output and volemia assessed by cardiac ultrasound, venous saturation in Oxygen (ScVO2) or ΔPP
* Hemodynamic stabilization : stable norepinephrine dosage (or <20% variations) with no vascular filling during the last 3 hours
* AKI stage I or II in KDIGO classification

Exclusion Criteria:

* Chronic Kidney Disease with glomerular filtration rate ≤ 30 ml/mn/1,73m2
* Obstructive AKI
* AKI stage III in KDIGO classification
* Known allergy to loop diuretics
* Contraindications to Furosemide
* FST not feasible within 12 hours of eligibility
* Previous AKI during the same hospitalization
* Pregnancy or breastfeeding women
* Subject under a legal protective measure
* No affiliation to a social regime or CMU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Need for renal replacement therapy or death | Before day 7
  Need for renal replacement therapy will be define according to the AKIKI study (Gaudry S, Hajage D, Schortgen F, Martin-Lefevre L, Pons B, Boulet E, et al. Initiation Strategies for Renal-Replacement Therapy in the Intensive Care Unit. N Engl J Med. 2016 Jul 14;375(2):122-33). Need for RRT following AKIKI delayed initiation criteria.
  FST performance will be compared to the need of RRT or death.
sensitivity | 3 hour after FST
  FST will be positive if patient is non responder : 2-hour urine output < 200mL

SECONDARY OUTCOMES:
6 hour urine output | 6 hour after FST
  measurement of urine out
percentage of effective renal replacement therapy | daily up to day 7
  Initiation of RRT
death | daily up to day 7
hemodynamic safety: noradrenaline dose | 6 hour after FST
  noradrenaline dose
clinical safety: arterial pressure | 6 hour after FST
  modification of systolic, diastolic or mean arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Cote Basque, Bayonne
  - Hopital Saint Louis, Paris
  - Hopital Bichat, Paris

IPD SHARING:
Plan to Share IPD: Undecided